CLINICAL TRIAL: NCT04296955
Title: Testing the Effect of a New Health Communication Intervention for Renal Transplant Recipients (KnowMAP).
Brief Title: Testing the Effect of KnowMAP (Knowledge Management for Renal Transplant Recipients). A Randomized Controlled Study
Acronym: KnowMAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Tone Vidnes, PhD student, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29385
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplantation
Keywords: health literacy; motivational interview; adherence; organ transplantation
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Interventional study model: Parallel assignment. 2- arm un-blinded RCT design. The arms are:
  1. The intervention: 4 individual patient counseling sessions using adapted motivational interviewing techniques in addition to usual care.
  2. Usual care: patients undergo standard patient education program for renal transplant recipients at OUS.
Masking Description: Block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health communication intervention (Experimental): Motivational interview as a new health communication intervention (one arm)
  Interventions: Other: Motivational interview as a new health communication intervention
- Standard care (No Intervention): Standard care

INTERVENTIONS:
Other: Motivational interview as a new health communication intervention — Same as intervention name
  Arms: Health communication intervention

SUMMARY:
A randomized controlled study (RCT) aiming to test the effect of a new health literacy intervention for renal transplant recipients, KnowMAP (knowledge management for renal transplant recipients).

DETAILED DESCRIPTION:
Every year about 250-300 kidney transplantations are performed at Oslo University Hospital in Norway. Considerable improvements have recently emerged within kidney transplantation in relation to survival and quality of life. However, after transplantation, adherence to immunosuppressive drug therapy and other medical advices is crucial for staying healthy, keeping the graft, and retain good quality of life. In case of graft loss the patient has to return to dialysis, representing reduced functioning, fatigue and negative impact on quality of life. Dialysis also leads to higher costs for the society and in many cases a need for re-transplantation. A key challenge to adherence is the ability to gain access to, understand and use health information, defined as health literacy by the WHO. For renal transplant recipients preparedness for handling information and going through transplantation is essential. Hence, supporting the patients becoming reflective and health literate knowledge users is crucial.

Through a RCT this project aims to test the effect of a new health communication intervention, KnowMAP (knowledge management for renal transplant recipients), as compared with standard care in patients undergoing renal transplantation.

KnowMap is a novel intervention designed by clinicians and researchers at Oslo University Hospital (OUS), University of Oslo (UiO) and University of Stavanger (UiS). The intervention is targeting knowledge management skills of patients by using motivational interview (MI) techniques. It represents 4 sessions of individual patient counselling starting the first week after the transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplanted patients > 18 years included within few days after kidney transplantation at Oslo University Hospital
* Able to speak and understand Norwegian

Exclusion Criteria:

* Not able to speak or understand Norwegian well enough to be able to fill out forms or have a conversation in Norwegian.
* Kidney transplanted patient <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Health literacy (HL) | 24 months post transplantation
  HL measured by the HLQ (Health Literacy Questionnaire): The HLQ includes 44 items over nine independent scales, each representing a different element of the overall HL construct. Each scale includes 4-6 items. The first five scales comprise items asking the respondents to indicate level of agreement [ranging from strongly disagree to strongly agree (range 1-4)]. The remaining scales (6-9) have domains of self-reported capability (range 1-5: 'cannot do' to 'very easy'). The questionnaire has no total score, as that could potentially mask individual needs in specific HL domains. The HLQ appears robust for its intended purpose of assessing HL in a range of settings and has shown excellent reliability.
Adherence to immunosuppressive medication | 24 months post transplantation
  The instrument BAASIS (The BAsel Adherence to immunoSuppressIve medication Scale) a self reporting adherence questionnaire measuring patients' taking, skipping, timing (>2 hrs from prescribed time) and dose reduction of drugs. The recall period is limited to four weeks. The BAASIS comprises four questions with a 6-point scale for responses ranging from never (0) to every day (5)

SECONDARY OUTCOMES:
Quality of life and cost-effectiveness estimates relevant to this clinical context | 24 months post transplantation
  using EQ-5D-5L, introduced by EuroQoL in 2009. It is a two pages, standardized generic questionnaire.
Knowledge | 24 months post transplantation
  Using a Norwegian developed questionnaire: "The Transplantation Knowledge Questionnaire"
Occations of graft loss | 24 months post transplantation
  Registred in the Norwegian Renal Registry (NNR)

CONTACTS AND LOCATIONS:
Overall Officials: Andersen, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway